CLINICAL TRIAL: NCT01399125
Title: A 24-Week, Randomized, Double-blind, Double-dummy, Parallel-group, Active-controlled Study to Assess the Efficacy, Safety, and Tolerability of the Once-daily Rivastigmine Patch Formulation in Patients With Probable Alzheimer's Disease (Mini-Mental State Examination (MMSE) 10-20)
Brief Title: A 24-Week Efficacy, Safety and Tolerability of Rivastigmine Patch Study in Patients With Probable Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CENA713D2344
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; Rivastigmine; Patch; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rivastigmine patch (Experimental): Once-daily target patch size 10 cm²
  Interventions: Drug: Rivastigmine Patch; Drug: Placebo to Rivastigmine capsules
- Rivastigmine capsules (Active Comparator): Twice-daily target dose of 6 mg oral capsule
  Interventions: Drug: Rivastigmine Capsules; Drug: Placebo to Rivastigmine patch

INTERVENTIONS:
Drug: Rivastigmine Patch — Once-daily target patch size 10 cm²
  Other Names: ENA713, Exelon
  Arms: Rivastigmine patch
Drug: Rivastigmine Capsules — Twice-daily target dose of 6 mg oral capsule
  Other Names: ENA713, Exelon
  Arms: Rivastigmine capsules
Drug: Placebo to Rivastigmine patch — Matching placebo to Rivastigmine patch
  Other Names: placebo
  Arms: Rivastigmine capsules
Drug: Placebo to Rivastigmine capsules — matching Placebo to Rivastigmine capsules
  Other Names: placebo
  Arms: Rivastigmine patch

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and tolerability of Exelon® patch in patients with probable AD (MMSE 10-20), in order to support a planned regulatory submission and registration of Exelon transdermal patch in China. The study is designed to confirm the non-inferiority of the efficacy of Exelon patch (target 10 cm² patch size) versus Exelon capsules (target 6.0 mg bid dose) on cognition, using the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog).

ELIGIBILITY:
Inclusion criteria:

* have a diagnosis of dementia of the Alzheimer's type according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria;
* have a clinical diagnosis of probable AD according to NINCDS/ADRDA criteria.
* have a brain scan (magnetic resonance imaging (MRI) or computed tomography (CT)) consistent with the diagnosis of AD. The brain scan must have been performed within one year prior to randomization;
* have an MMSE score of ≥ 10 and ≤ 20;
* have sufficient education to have been able to read, write, and communicate effectively during the premorbid state;
* be residing with someone in the community throughout the study or, if living alone, in contact with the primary caregiver everyday;

Exclusion criteria:

* have an advanced, severe, progressive, or unstable infectious, metabolic, immune, endocrinologic, hepatic, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological condition that may interfere with efficacy and safety assessments or put the patient at special risk;
* have a history or current diagnosis of any medical or neurological condition other than AD that is identified as contributing cause of the patient's dementia;
* have a current diagnosis of probable or possible vascular dementia according to the National Institute of Neurological Disorders and Stroke and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences criteria (NINDS-AIREN);
* have a score of > 4 on the Modified Hachinski Ischemic Scale (MHIS);
* have a current DSM-IV diagnosis of major depression, unless, in the opinion of the investigator, is in remission for at least 12 weeks;

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- China (11):
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rivastigmine Patch | Rivastigmine Capsules
Started | 248 | 253
Per Protocol (PP) Population | 192 | 188
Completed | 197 | 193
Not Completed | 51 | 60
Not completed — Adverse Event | 32 | 30
Not completed — Abnormal Lab values | 0 | 1
Not completed — Unsatisfactory Therapeutic Effect | 0 | 4
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Lost to Follow-up | 2 | 3
Not completed — Administrative Problems | 7 | 11
Not completed — Death | 0 | 1
Not completed — Protocol Deviation | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivastigmine Patch | Rivastigmine Capsules | Total
Number analyzed (Participants) | 248 | 253 | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (8.02) | 69.8 (8.20) | 70.1 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 139 | 279
  Male | 108 | 114 | 222

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Cognition, Assessed by the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog)
Description: The Alzheimer's Disease Assessment Scale (ADAS) is a performance-based test that measures specific cognitive and behavioral dysfunctions in patients with Alzheimer's Disease. The cognitive subscale of the ADAS (ADAS-Cog) comprises 11 items that are summed to a total score ranging from 0 to 70, with lower scores indicating less severe impairment. It was assessed by a mental health professional (e.g., M.D., Ph.D., Pharm.D., R.N., or other equivalent qualifications) with a minimum of 2 years research experience meeting certification requirements.
Time Frame: Change at 24 weeks
Population: Per Protocol (PP): patients who received at least one dose of study drug, had a baseline assessment and at least one post-baseline assessment on treatment (after Day 140 and not more than 2 days after the last known date of study drug) of the primary efficacy variable and have no major protocol deviations.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rivastigmine Patch | Rivastigmine Capsules
Number analyzed (Participants) | 192 | 188
Scores on a scale | -0.5 (6.70) | -0.7 (6.74)

2. Secondary Outcome: Change From Baseline in Global Functioning, Assessed by the Alzheimer's Disease Assessment Scale Clinical Impression of Change (ADCS-CGIC)
Description: Alzheimer's disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) scale provides a single global rating of change from baseline. It was recommended that the baseline interview be conducted by two raters, one designated as the primary rater, the other as a backup. Both raters were independent trained clinicians, experienced in the assessment of patients with dementia. Neither rater was involved in any other way with the patients' treatment or evaluation throughout the study. At baseline, both raters had access to all of the patient's available records and evaluations. Subsequently, for all ratings of change from baseline, the rater relied solely on information obtained during the baseline interview of the patient and caregiver, including written notes and, if available, the baseline interview audio- or videotape. The rater had no access to any other safety or efficacy data, including all previous post-baseline ADCS-CGIC ratings by either rater.
Time Frame: Change at 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Rivastigmine Patch | Rivastigmine Capsules
Number analyzed (Participants) | 192 | 188
participants
  marked improvement | 1 | 1
  Moderate improvement | 10 | 12
  Minimal improvement | 68 | 59
  No change | 67 | 74
  Minimal worsening | 38 | 35
  Moderate worsening | 7 | 6
  Marked worsening | 1 | 0

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) Total Score
Description: Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) is a caregiver-based Activities of Daily Living (ADL) scale composed of 23 items developed for use in dementia clinical studies. It was designed to assess the patient's performance of both basic and instrumental activities of daily living such as those necessary for personal care, communicating and interacting with other people, maintaining a household, conducting hobbies and interests, as well as making judgments and decisions. Responses for each item were obtained from the caregiver through an interview. For each basic ADL, there was a forced choice of best response or a "yes" or "no" question with additional sub questions. Higher numbered scores and answers of "yes" reflected a more self-sufficient individual. Therefore, the higher total score, the higher functioning the patient was. The total score was the sum of all items and sub questions. The range for the total ADCS-ADL score was 0 to 78.
Time Frame: Change at 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch | Rivastigmine Capsules
Number analyzed (Participants) | 192 | 188
scores on a scale | -1.9 (11.02) | -1.7 (11.31)

4. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score
Description: NPI including Caregiver Distress Scale (NPI-D) assesses a wide range of behavior problems encountered in dementia patients to provide a means of distinguishing frequency and severity of changes in behavioral problems & facilitates rapid behavioral assessment using screening questions.10 behavioral problems & 2 neurovegetative domains were evaluated through an interview of the caregiver by a mental health professional. The scale includes both frequency & severity ratings of ea. domain as well as a composite domain score(frequency x severity). Frequency: 1(occasionally) - 4(very frequently)&severity:1(mild) - 3(marked).The sum of the composite scores of the 12 domains yields the NPI total score. The NPI-D: 0(not severe & not at all distressing) - 5 (very severe or extremely distressing) for each of the 12 domains. NPI-12 total score: from 0-144, the NPI-10 total score: from 0-120, & NPI-D score: from 0-60, all with higher scores indicating more severe behavioral disturbance.
Time Frame: Change at 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch | Rivastigmine Capsules
Number analyzed (Participants) | 192 | 188
scores on a scale
  NPI-12: Total score (frequency x severity) | -1.3 (11.22) | -1.3 (11.98)
  NPI-10: Total score (frequency x severity) | -1.2 (9.84) | -1.3 (10.46)
  NPI-D: Distress score (frequency x severity) | -0.4 (5.65) | -0.6 (5.88)

5. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Total Score
Description: The Mini-Mental State Examination (MMSE) was used to establish patient's eligibility for the study and it was also used as an efficacy parameter in the Double-blind Treatment Period. The MMSE is a brief, practical screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language) and results in a total possible score of 30, with higher scores indicating betterfunction. The total MMSE score at screening was between 10 and 20, inclusive, in order forthe patient to be eligible to participate in the trial.
Time Frame: Change at 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch | Rivastigmine Capsules
Number analyzed (Participants) | 192 | 188
scores on a scale | 0.7 (3.31) | 0.7 (3.30)

ADVERSE EVENTS:
Description: In participant Flow 248 patients (Rivastigmine Patch) and 253 patients (Rivastigmine Capsules) were randomized. For the Adverse Events the Safety (SAF) population: patients who received at least one dose of study drug, and had at least one post-baseline safety assessment was analyzed there fore 247 and 251 patients respectively
Groups:
- Rivastigmine Capsule: Twice-daily target dose of 6 mg oral capsule
Arm/Group | Rivastigmine Patch | Rivastigmine Capsule
Serious Adverse Events (participants affected / at risk) | 16/247 | 21/251
Other Adverse Events (participants affected / at risk) | 82/247 | 111/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Patch (N=247) | Rivastigmine Capsule (N=251)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Diabetic coma (Nervous system disorders) | 1 | 0
Anorexia nervosa (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Patch (N=247) | Rivastigmine Capsule (N=251)
Diarrhoea (Gastrointestinal disorders) | 5 | 8
Nausea (Gastrointestinal disorders) | 20 | 32
Vomiting (Gastrointestinal disorders) | 19 | 31
Application site pruritus (General disorders) | 27 | 7
Medication error (Injury, poisoning and procedural complications) | 10 | 7
Weight decreased (Investigations) | 10 | 17
Decreased appetite (Metabolism and nutrition disorders) | 16 | 37
Dizziness (Nervous system disorders) | 15 | 25
Somnolence (Nervous system disorders) | 6 | 11
Insomnia (Psychiatric disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.